CLINICAL TRIAL: NCT05371249
Title: Seven-Day Vonoprazan-Based Triple Therapy With High-Dose Amoxicillin as First-Line Helicobacter Pylori Treatment in Comparison With Extended Sequential Therapy: A Randomized Controlled Trial in Taiwan
Brief Title: Vonoprazan-Based Triple Therapy in Comparison With Extended Sequential Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJUH110108
Record Dates: First submitted 2022-04-24; First posted 2022-05-12 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Helicobacter Pylori
Keywords: Proton Pump Inhibitors
MeSH Terms: interventions — ribosomal protein S14

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan-based triple therapy group (Experimental): Including patients receiving vonoprazan-based triple therapy (vonoprazan 20mg + amoxicillin 1000 mg + clarithromycin 500 mg twice daily for seven days)
  Interventions: Drug: Vonoprazan-based triple therapy
- Extended sequential therapy group (Active Comparator): Including patients receiving extended sequential therapy (lansoprazole 30mg + amoxicillin 1000mg twice daily for 7 days, followed by lansoprazole 30mg + clarithromycin 500mg + metronidazole 500mg twice daily for 7 days)
  Interventions: Drug: Extended sequential therapy

INTERVENTIONS:
Drug: Vonoprazan-based triple therapy — vonoprazan 20mg+amoxicillin 1000 mg + clarithromycin 500 mg twice daily for seven days
  Other Names: VAC-7
  Arms: Vonoprazan-based triple therapy group
Drug: Extended sequential therapy — Lansoprazole 30mg + amoxicillin 1000mg twice daily for 7 days, followed by lansoprazole 30mg + clarithromycin 500mg + metronidazole 500mg twice daily for 7 days
  Other Names: S-14
  Arms: Extended sequential therapy group

SUMMARY:
This study aims to compare the efficacy of the current standard first-line anti-helicobacter pylori regimen, extended proton pump inhibitor-based sequential therapy, with that of vonoprazan-based triple therapy, through a randomized controlled trial.

DETAILED DESCRIPTION:
Helicobacter pylori infection is a well-established risk factor for peptic ulcer disease and gastric cancer. It's now a consensus of experts that H.pylori infection should be treated once it is recognized. Extended proton pump inhibitor (PPI)-based sequential therapy as one of the most commonly used first-line regimens provides a satisfactory eradication rate of 90.7% (95% CI, 87.4% - 94.0%). Nevertheless, its complexity of the "sequential" usage is sometimes confusing to the patients and may lead to treatment failure. The emerging new regimen - vonoprazan-based triple therapy, on the other hand, is another appealing choice with simplicity, short treatment duration, and low pill burden. However, there's still no evidence regarding the use of vonoprazan-based triple therapy with high-dose amoxicillin (1000mg twice daily) as the first-line regimen. This study aimed to compare the efficacy of the current standard first-line regimen, sequential therapy, with that of vonoprazan-based triple therapy with high-dose Amoxicillin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with H.pylori infection who was over 20 years old and agree to participate in the trial will be recruited.

Exclusion Criteria:

* Who had received helicobacter pylori eradication before
* Who are known to be allergic to any drug used in this trial
* Pregnant women
* Who are refuse to participate in the trial for any reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of helicobacter pylori | Assessed at least 6 weeks after the therapy
  Assessed by urea breath test

SECONDARY OUTCOMES:
Adverse effects of the drugs | After patients completed the therapy (For VAC-7 group: 1 week after the therapy; For S-14 group: 2 weeks after the therapy)
  Self-reported adverse effects by patients through a questionnaire.
Compliance | After patients completed the therapy ((For VAC-7 group: 1 week after the therapy; For S-14 group: 2 weeks after the therapy)
  Self-reported compliance by patients through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-tse Chiu, MD, Study Chair — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study will be stored in a non-publically available repository and are available on request for the use of academic research in relevant field after the study is published, in the form of excel file with de-identification (main contact: Chiu, Yu-tse, b95401030@gmail.com; consent from participants had been obtained).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available on request for the use of academic research in relevant field after the study is published.
Access Criteria: The purpose of obtaining the IPD should be for the use of academic research in relevant field.

REFERENCES:
- [Derived] Chiu YT, Lee FJ, Kuo CY, Chen YT, Lin YC, Liang KS, Wu CY, Lin RT, Lin JT, Chang CY. Seven-Day Vonoprazan-Based Triple Therapy as First-Line Helicobacter pylori Treatment in Comparison With Extended Sequential Therapy: A Randomized Controlled Trial. Helicobacter. 2024 Jul-Aug;29(4):e13129. doi: 10.1111/hel.13129. PMID 39164808